CLINICAL TRIAL: NCT05498987
Title: Ultrasound Achilles Tendon Assessment After 448kilohertz Capacitive Resistive Radiofrequency Stimulation in a Sporty Population
Brief Title: Ultrasound Achilles Tendon Assessment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, María Cuevas Cervera, Principal Investigator, Universidad de Granada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCuevasCervera
Record Dates: First submitted 2022-07-17; First posted 2022-08-12 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Ultrasonography; Achilles Tendon

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 448 kilohertz Capacitive Resistive Monopolar Radiofrequency stimulus on the dominant Achilles Tendon (Experimental): 448 kilohertz Capacitive Resistive Monopolar Radiofrequency stimulus on the dominant Achilles Tendon
  Interventions: Device: Monopolar 448 kilohertz radiofrequency stimulation

INTERVENTIONS:
Device: Monopolar 448 kilohertz radiofrequency stimulation — 448kilohertz capacitive resistive monopolar radiofrequency will be applied on the dominant Achilles Tendon

SUMMARY:
448kilohertz capacitive resistive monopolar radiofrequency is a novel technique in physiotherapy and its usefulness and clinical relevance is still to be investigated at both clinical practice and also in performance. Current studies show promising results in different musculoskeletal disorders, however there no studies in the assessment of quality soft tissue in sporty population after the used of this technique.

DETAILED DESCRIPTION:
Achilles Tendon pain is is one of the most common musculoskeletal disorders, presenting a high prevalence in primary care centers and sport populations. Many factors have been proposed as the cause of pain, however there are no studies analysing possibilities of preventing Achilles Tendon injuries by using a radiofrequency stimulus.

The use of 448kilohertz capacitive resistive monopolar radiofrequency as the focus of the treatment looking for improve the quality of the tissue is still to be explored.

The hypothesis of the present project is that focus treatments on 448kilohertz capacitive resistive monopolar radiofrequency on the Achilles Tendon will produce better outcomes in terms of ultrasound assessment measured by quantified elastography, and this will decreased the possibilities of get injured.

The stimulus will be carried out on the Achilles Tendon region. All interventions will be developed by the same examiner, who is a physiotherapist with 6 years of clinical experience.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-50 years
* Sporty people with at least 3 days of training per week and presenting an upper limb dominance.

Exclusion Criteria:

* Suffer from any painful Achilles Tendon condition.
* History of significant Achilles Tendon trauma, such as fracture or ultrasonography Clinically suspected partial thickness cuff tear, following the classification of Wiener and Seitz.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-05-14 (Estimated); Primary Completion 2023-06-14 (Estimated); Study Completion 2024-06-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Achilles Tendon measured by quantified elastography imaging at 3 months. time (t) 1(prior to treatment), t2 (immediately after the treatment), t3 (3 months later). | time (t) 1(prior to treatment), t2 (immediately after the treatment), t3 (3 months later). Changes in tendinous thickness [ Time Frame: 9 months ]
  The elastography is obtained when the anatomic image on grayscale ultrasound overlaps parametric color image that expresses the rate of deformity of the tissues, soft tissues tend to develop greater deformity and tissue deformity have lower rigidity.

CONTACTS AND LOCATIONS:
Locations (1):
- Ana Gonzalez Muñoz, Málaga, Malaga, Spain